CLINICAL TRIAL: NCT03267771
Title: Role of Serum Progesterone and Doppler Ultrasound in Prediction of Pregnancy Outcome in Women With Recurrent Unexplained Abortion
Brief Title: Progesterone and Doppler in Recurrent Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, GKElsherief, prinicipal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gehad elsherief
Record Dates: First submitted 2017-06-05; First posted 2017-08-30 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Abortion in First Trimester
MeSH Terms: interventions — Dydrogesterone; Ultrasonography, Doppler

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- progesterone suppositories vaginal group (Active Comparator): vaginal micronized progesterone suppositories (prontogest®) 400 mg, one vaginal suppository twice daily through 18 weeks of gestation.
  Interventions: Drug: Progesterone Suppositories Vaginal; Device: doppler ultrasound
- Dydrogesterone oral tablets group (Experimental): 20 mg tablets (Duphaston ®), 2 tablets orally twice daily through 18 weeks of gestation.
  Interventions: Drug: Dydrogesterone Oral Tablet; Device: doppler ultrasound

INTERVENTIONS:
Drug: Progesterone Suppositories Vaginal — progesterone vaginal suppository
  Other Names: Prontogest
  Arms: progesterone suppositories vaginal group
Drug: Dydrogesterone Oral Tablet — oral progesterone drug
  Other Names: Duphaston
  Arms: Dydrogesterone oral tablets group
Device: doppler ultrasound — pulsed doppler ultrasound
  Other Names: Gomez et al

SUMMARY:
Recurrent pregnancy loss is classically defined as the occurrence of three or more consecutive pregnancy loss. The American Society of Reproductive Medicine has recently redefined recurrent pregnancy loss as two or more pregnancy losses. A pregnancy loss is defined as a clinically-recognized pregnancy means that the pregnancy has been visualized on an ultrasound or that pregnancy tissue was identified after a pregnancy loss.

DETAILED DESCRIPTION:
Spontaneous pregnancy loss is a surprisingly common occurrence. Whereas approximately 15% of all clinically recognized pregnancies result in spontaneous loss, there are many more pregnancies that fail prior to being clinically recognized. Only 30% of all conceptions result in a live birth.

Although no reliable published data have estimated the probability of finding an etiology for recurrent pregnancy loss in a population with 2 versus 3 or more miscarriages, the best available data suggest that the risk of miscarriage in subsequent pregnancies is 30% after 2 losses, compared with 33% after 3 losses among patients without a history of a live birth. This strongly suggests a role for evaluation after just 2 losses in patients with no prior live births. An earlier evaluation may be further indicated if fetal cardiac activity was identified prior to a loss .

ELIGIBILITY:
Inclusion Criteria:

1. pregnant 7-12 weeks documented by pregnancy test &/or ultrasaound.
2. History of at least 2 prior spontaneous abortion before 12 weeks of gestation.
3. Age: 18-35 years
4. Willing and able to give informed consent.
5. Rh +ve patient
6. BMI: 18-32
7. Viable pregnancy through the detection of fetal pulsations by ultrasound
8. Singleton pregnancy
9. Apparently stable pregnancy (no history of vaginal bleeding in this current pregnancy or signs of sac separation in ultrasound)

Exclusion Criteria:

1. Patients diagnosed to have Anti-phospholipid syndrome or another recognised thrombophilic or autoimmune conditions.
2. Pregnant > 12 weeks.
3. Contraindication to progesterone use.
4. Diabetic patients, have glucose intolerance.
5. Multiple pregnancies.
6. Thyroid disorder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-08-05 (Estimated); Study Completion 2019-12-05 (Estimated)

PRIMARY OUTCOMES:
number of Live births after 28 weeks of gestation | 28 weeks gestation
  Live births that survive and continue beyond 28 weeks of gestation

SECONDARY OUTCOMES:
Number of patients who Tolerable with the treatment | 12 weeks
  efficacy of treatment on patients

CONTACTS AND LOCATIONS:
Locations (1):
- Gehad Elsherief, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macklon NS, Geraedts JP, Fauser BC. Conception to ongoing pregnancy: the 'black box' of early pregnancy loss. Hum Reprod Update. 2002 Jul-Aug;8(4):333-43. doi: 10.1093/humupd/8.4.333. PMID 12206468
- [Background] Sotiriadis A, Papatheodorou S, Makrydimas G. Threatened miscarriage: evaluation and management. BMJ. 2004 Jul 17;329(7458):152-5. doi: 10.1136/bmj.329.7458.152. No abstract available. PMID 15258071